CLINICAL TRIAL: NCT03357081
Title: Utility of Real-Time Contrast Enhanced Ultrasound (CEUS) in the Evaluation of Soft Tissue Hematomas
Acronym: CEUS
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Tobias Kummer, Principle Investigator, Mayo Clinic
Other Study IDs: 17-004506
Record Dates: First submitted 2017-09-19; First posted 2017-11-29 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Hematoma
MeSH Terms: conditions — Hematoma | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- CEUS: Adult patients over the age of 18 who have a clinical suspicion of an actively bleeding soft-tissue hematoma as determined by the treating emergency provider. Enrollment will be for one year or until a target of 20 patients is enrolled.
  Interventions: Drug: CEUS or Contrast enhanced Ultrasound

INTERVENTIONS:
Drug: CEUS or Contrast enhanced Ultrasound — Real time contrast enhanced ultrasound with Lumason. CEUS or Contrast enhanced Ultrasound
  Other Names: Ultrasound; CEUS with Lumason

SUMMARY:
Traumatic and non-traumatic soft tissue hematomas are frequently encountered in the acute care setting. The incidence of these hematomas appears to be on the rise secondary to the increased use of anticoagulants among older patients for a variety of medical conditions.

The management of soft tissue hematomas depends on the accurate diagnosis of any ongoing bleeding as well as of identification of the injured vessel type. While the majority of cases can be managed conservatively, expanding hematomas leading to hemodynamic instability or ongoing blood loss might require embolization or surgical intervention. The mainstay diagnostic imaging modality is multidetector computed tomography (MDCT) with intravenous contrast that allows accurate assessment of hematoma size, location as well as evaluation for active extravasation. However, many patients cannot undergo CT imaging due to underlying kidney disease, allergy to contrast, or due to concerns for radiation exposure, especially in young age. Currently there are no alternative tests for these patients with a similarly high diagnostic accuracy available.

This study intends to establish an imaging protocol and investigate the utility of contrast-enhanced ultrasound (CEUS) in the diagnostic work-up of soft tissue hematoma as an ionizing radiation-free alternative to computed tomography (CT) that can be used independent from the kidney function of the patient.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over the age of 18 who have a clinical suspicion of an actively bleeding soft-tissue hematoma as determined by the treating emergency provider. Enrollment will be for one year or until a target of 20 patients is enrolled.

Exclusion Criteria:

* The investigators will exclude persons under the age of eighteen, vulnerable populations (pregnant patients and prisoners), need for immediate procedural intervention and those with known hypersensitivity to sulfur hexafluoride lipid containing microspheres as well as those who have a soft-tissue hematomas that are in an unfavorable anatomical location for ultrasound imaging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patient's will be enrolled during the partcipants Emergency Department evaluation at St. Mary's Hospital, Rochester, MN.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2019-09-22 (Actual); Study Completion 2019-09-22 (Actual)

PRIMARY OUTCOMES:
Contrast-pooling within the hematoma as a sign of active extravasation | 1 year
  Contrast outside of the blood vessel indicates ongoing bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Kummer, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
This pilot study will allow us to develop ultrasound scanning parameters and protocols. Successful preliminary data of this pilot study would allow our team to apply for extramural funding for a larger clinical trial to assess the diagnostic accuracy of CEUS in the evaluation of these hematomas

REFERENCES:
- [Derived] Kummer T, Mohn KJ, Bardwell AJ, Boyum JH. Evaluation of Soft-Tissue Hematomas With Real-Time, Contrast-Enhanced Ultrasound: A Pilot Study With Preliminary Findings. Ultrasound Q. 2023 Sep 1;39(3):179-185. doi: 10.1097/RUQ.0000000000000621. PMID 36731072
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials